CLINICAL TRIAL: NCT04338997
Title: An Open-label Phase 1b Study to Evaluate the Pharmacokinetics and Pharmacodynamics in Plasma and Cerebrospinal Fluid (CSF), Safety and Tolerability of Oral IZD174 in Patients With Parkinson's Disease
Brief Title: PK Study in Patients With Parkinson's Disease With IZD174
Status: Withdrawn | Phase: Phase 1 | Type: Interventional
Why Stopped: Strategic decision by Sponsor
Sponsor: Inflazome UK Ltd (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: IZD174-003
Record Dates: First submitted 2020-04-03; First posted 2020-04-08 (Actual); Last update posted 2020-12-04 (Actual); Status verified 2020-09

CONDITIONS: Parkinson Disease
MeSH Terms: conditions — Parkinson Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- IZD174 (Experimental): Intra subject dose escalation of IZD174
  Interventions: Drug: IZD174

INTERVENTIONS:
Drug: IZD174 — Small molecule inhibitor of NLRP3

SUMMARY:
Single center, open-label, intra-individual dose-escalation study in subjects with mild/moderate Parkinson's Disease

DETAILED DESCRIPTION:
After assessing eligibility during a screening period of up to 4 weeks, up to 6 subjects will be included.

Subjects will check into the clinic one day prior to dosing (Day -1). To evaluate and compare drug exposure levels in plasma and CSF, plasma and CSF will be serially sampled over a period of 36 hours. Subjects will be discharged from the clinic on Day 5 after all required study procedures are completed and if medically justified.

Subjects will return to the clinic approximately 1 week after discharge from the clinic for a follow-up visit.

ELIGIBILITY:
Inclusion Criteria:

* The subject is a man or woman aged between 45 and 75, inclusive.
* Documented clinically established diagnosis of Parkinson's Disease, Hoehn & Yahr stage 1 to 3 and Montreal Cognitive Assessment greater or equal than 26. Diagnosis of Parkinson's Disease consistent wit MDS Research Criteria for the Diagnosis of Parkinson's Disease must include bradykinesia with sequence effect, and motor asymmetry (especially if no rest tremor). Diagnosis has to be made less than 3 years prior to Screening.
* The subject understands the nature and purpose of the study, including possible risks and side effects, and i willing and able to comply with all compulsory stud procedures and provides signed and dated written informed consent (in accordance with local regulations) prior to any study procedures being performed.

Exclusion Criteria:

* The subject used any NSAIDs, steroids, colchicine or anti-IL-1 inhibitors within 7 days prior to Day 1.
* The subject received any investigational drugs within 4 weeks or 5 half-lives (whichever is longer), prior to Day 1.
* The subject had an active systemic infection (other than common cold) within 2 weeks prior to Day 1.
* The subject has a history of severe hypersensitivity to previous drugs.
* The subject has any severe, progressive or uncontrolled medical condition at Screening or on Day -1 that in the judgment of the investigator prevents the subject from participating in the study.

Ages: 45 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2020-10 (Estimated); Primary Completion 2020-11 (Estimated); Study Completion 2020-12 (Estimated)

PRIMARY OUTCOMES:
Concentration of IZD174 in plasma | Pre-dose to 36 hours post dose
  Plasma PK profile following an intra-individual dose escalation of IZD174
Concentration of IZD174 in cerebrospinal fluid | Pre-dose to 36 hours post dose
  CSF PK profile following an intra-individual dose escalation of IZD174
Ratio of IZD174 concentration in plasma to CSF | Pre-dose to 36 hours post dose
  CSF to plasma concentration ratio at each time point

SECONDARY OUTCOMES:
Inhibition of Interleukin-1 beta secretion in ex-vivo stimulated whole blood | Pre-dose to 36 hours post dose
  Inhibition of IL-1 secretion by ex-vivo stimulated whole blood
Incidence of Treatment-Emergent Adverse Events | Day 0 to Day 10
  Safety & Tolerability as measured by incidence if Treatment-Emergent Adverse events

CONTACTS AND LOCATIONS:
Overall Officials: Teus van Laar, MD, PhD, Principal Investigator — UMCG Groningen

IPD SHARING:
Plan to Share IPD: No